CLINICAL TRIAL: NCT07056439
Title: A Phase I/II Clinical Study to Evaluate the Safety, Pharmacokinetics, Radiation Dosimetry and Preliminary Diagnostic Efficacy of HRS-1738 in PET/CT Imaging of Patients With Prostate Cancer
Brief Title: Phase I/II Clinical Study of HRS-1738 for the Diagnosis of Prostate Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HRS-1738-101
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: PET Imaging in Patients With Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-1738 Group (Experimental)
  Interventions: Drug: HRS-1738 Injection

INTERVENTIONS:
Drug: HRS-1738 Injection — HRS-1738 injection.

SUMMARY:
This study aims to evaluate the safety and pharmacokinetics of HRS-1738 injection in adult patients with prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and abide by the procedures and requirements of this study and voluntarily sign the informed consent form.
2. Male, aged ≥18 years old.
3. ECOG (Eastern Oncology Collaboration) Physical Condition score: 0 or 1.
4. Prostate adenocarcinoma confirmed by histopathology.
5. The distance between enrollment and the most recent surgical treatment should be at least 12 weeks. If the patient has recovered from the surgery before enrollment and meets other enrollment criteria, it can be relaxed to 8 weeks as determined by the investigator.
6. The functions of the major organs should meet the requirements.
7. For male subjects, they need to agree to take effective contraceptive measures with their partners within one week after the last administration of the investigational drug from the date of signing the informed consent form, and have no plans for fertility and do not donate sperm.

Exclusion Criteria:

1. Combined with the following diseases:

   1. . Severe urinary incontinence, hydronephrosis, severe urinary dysfunction, etc. Note: Subjects with bladder outflow tract obstruction or urinary incontinence who can be controlled through the existing best standard treatment (including urinary pads, drainage, etc.) are eligible to participate in the study.
   2. . Concurrent active infection or unexplained fever >38.5℃ for more than 1 hour during the screening period and before administration.
   3. . Combined with severe or poorly controlled systemic diseases, including but not limited to poorly controlled diabetes, congestive heart failure, unstable angina pectoris, myocardial infarction that occurred within 6 months before administration, refractory hypertension, acute kidney injury, stroke, and severe liver injury.
   4. . Combined with active hepatitis B (HBV-DNA testing is required for HBsAg positive patients, and HBV DNA≥2000 IU/mL or 104 copies/mL), active hepatitis C (HCV-Ab positive and higher than the detection limit of the analytical method).
   5. . Those who are known to have tested positive for acquired immunodeficiency syndrome (AIDS) or human immunodeficiency virus (HIV).
   6. . Active syphilis infected individuals.
2. According to the NCI-CTCAE v5.0 classification, those whose toxicity caused by previous anti-tumor treatment has not yet recovered to grade ≤1 (except for decreased lymphocyte count alone, alopecia, and the indicators mentioned in the inclusion criteria; According to the judgment of the researchers, after consultation with the sponsor, some tolerable chronic grade 2 toxicities may be excluded.
3. There are any factors that prevent the smooth progress of PET/CT examination or interfere with the interpretation of imaging results, including but not limited to the following situations: such as inability to lie flat, remain still or tolerate PET/CT scanning; It is known that there are metal implants or joint prostheses, etc.
4. It is known that there is an allergy or contraindication to any component of the test drug or its preparation.
5. Patients who had a second primary malignant tumor other than prostate cancer before enrollment, excluding malignant tumors with a low risk of metastasis and death that have been cured (5-year survival rate >90%), such as superficial squamous cell carcinoma of the skin, low-grade superficial bladder cancer, etc.
6. History of neurological or mental disorders, including epilepsy or dementia.
7. Participating in other clinical studies or having less than 4 weeks since the end of the last administration of the previous clinical study at the time of the first administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | About 1 year.
Serious adverse events (SAEs) | About 1 year.

SECONDARY OUTCOMES:
The maximum blood drug concentration (Cmax) | About 1 year.
Time to peak (Tmax) | About 1 year.
Biological half-life (t1/2) | About 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided